CLINICAL TRIAL: NCT06086782
Title: Comparative Effects of Autogenic and Reciprocal Inhibition Techniques on Pain, Disability and Range of Motion Among Smart Phone User With Trapezitis
Brief Title: Effects of Autogenic and Reciprocal Inhibition on Trapezitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0145
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Neck Pain
Keywords: trapezitis; Disability; neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autogenic inhibition (Experimental): isometric of muscles and stretching of the same side
  Interventions: Other: autogenic inhibition
- reciprocal inhibition (Experimental): isometric of muscles and stretching of the opposite side
  Interventions: Other: reciprocal inhibition

INTERVENTIONS:
Other: autogenic inhibition — Group 1 will receive AI-MET with conventional treatment. AI include stretching of the affected muscle and performing isometric contraction with 50% of the total patient's effort in the same muscle that will being stretched and position hold for 10 seconds, with 5 seconds of rest after every repetition. This procedure will repeat 5 times.
  Arms: autogenic inhibition
Other: reciprocal inhibition — Group 2 receive RI-MET with conventional treatment. The RI also include stretching of the affected muscle but contrary to AI, isometric contraction of the antagonist muscles with the 50% of total patient's effort will follow. This position holds for 10 seconds, while agonist's muscle will still in the stretched position, with 5 seconds of rest after every repetition. This procedure will repeat 5 times too.
  Arms: reciprocal inhibition

SUMMARY:
Aim of my study is to compare two techniques of METS i.e., autogenic and reciprocal inhibition techniques on pain, disability and Range of motion among smart phone user with trapezitis.

DETAILED DESCRIPTION:
Study focuses trapezitis in smart phone users. There are many different causes of neck pain, but one common factor is upper trapezitis. This refers to pain and spasms in the neck caused by inflammation of the trapezius muscle. The aim of this study is to compare the effects of autogenic and reciprocal inhibition techniques on pain, range of motion and disability among smart phone user with trapezitis.

This study will be randomized clinical trial and 40 patients male and female with age 20 to 40 years having NPRS >3 according to inclusion criteria will be included in the study. They will be allocated into 2 groups by non-probability convenience sampling technique. Group A will receive autogenic inhibition technique with conventional physical therapy while Group B will receive reciprocal inhibition technique with conventional therapy. Outcome measures; Neck Disability Index, goniometry and Numeric Pain Rating Scale will measure neck function and neck pain intensity. Total 12 sessions, 3 sessions per week for 4 weeks were provided. Each session was 45 minutes long and measurements will be taken at the baseline and at the end of 4th week. Data will be analyzed by SPSS version 25

ELIGIBILITY:
Inclusion Criteria:

* Mobile phone users age between 20 -40 years old.
* Both gender male and female included.
* Neck pain (Numeric Pain Rating Scale >3)
* With limited Neck ROMs.
* NDI scoring 15-24points (30-48%) moderate disability

Exclusion Criteria:

* Neck pain with whiplash or headache, neurological disorder.
* History of previous head, neck, cervical spine or shoulder surgery.
* Infection or inflammatory arthritis in the cervical spine.
* Trigger point of Upper trapezius will be excluded.
* History of cervical radiculopathy.
* Diagnosed fibromyalgia and myopathy.
* History of cancer.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Goniometry | 4 weeks
  The art and science of measuring the joint ranges in each plane of the joint are called goniometry. The term 'goniometry' has its origin from two Greek words, gonia, which means angle, and metron, which means to measure. Goniometer is a device that measures an angle or permits the rotation of an object to a definite position. A universal goniometer has three parts. The fulcrum and the body are placed over the joint being measured. The stationary arm is the arm of the goniometer that aligns with the inactive part of the joint measured. It is structurally a part of the body and is not movable independently of the body. The moving arm is the arm of the goniometer, which aligns with the mobile part of the joint measured. Neck flexion, extension, side bending and rotation will be assessed through it

SECONDARY OUTCOMES:
NPRS (numeric pain rating scale) | 4 weeks
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a unidimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale. The common format is a horizontal bar or line. Although various iterations exist, the most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"). The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10) that best reflects the intensity of his/her pain 11-point numeric scale ranges from '0' representing no pain to 10 representing the worst imaginable pain. Reliability of NPRS is (r=0.96 and 0.95) and validity is from 0.86 to 0.95
NDI (neck disability index) | 4 weeks
  The Neck Disability Index (NDI) (modification of the Oswestry Low Back Pain Disability Index). This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life. The NDI has become a standard instrument for measuring self-rated disability due to neck pain. Each of the 10 items scores from 0 to 5. Scoring for each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. The maximum score is 50 (20). Reliability of NDI is 0.50 and 0.98

CONTACTS AND LOCATIONS:
Overall Officials: Humera Mubashar, MS, Principal Investigator — Riphah International University
Locations (1):
- Nusrat Rashid Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No